CLINICAL TRIAL: NCT03078257
Title: Different Platelet Activities Between Intracoronary and Peripheral Blood in Coronary Artery Disease Patients
Acronym: DPABIAP
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Chunjian Li, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 005
Record Dates: First submitted 2017-02-23; First posted 2017-03-13 (Actual); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Coronary Artery Disease
Keywords: Platelet Activities; light aggregometry; VerifyNow P2Y12-assay; peripheral vein; peripheral artery; intracoronary artery; tirofiban; antiplatelet thrombolysin
MeSH Terms: conditions — Coronary Artery Disease | interventions — Tirofiban; Clopidogrel; Aspirin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- dual antiplatelet therapy (Experimental): clopidogrel +aspirin
  Interventions: Drug: Clopidogrel; Drug: Aspirin
- tirofiban in PV (Experimental): clopidogrel +aspirin + tirofiban in PV
  Interventions: Drug: tirofiban in PV; Drug: Aspirin; Drug: Clopidogrel
- tirofiban in IC (Experimental): clopidogrel +aspirin +tirofiban in IC
  Interventions: Drug: tirofiban in IC; Drug: Aspirin; Drug: Clopidogrel
- antiplatelet thrombolysin (Experimental): clopidogrel +aspirin +antiplatelet thrombolysin
  Interventions: Drug: antiplatelet thrombolysin; Drug: Aspirin; Drug: Clopidogrel
- placebo (Placebo Comparator): clopidogrel +aspirin +placebo
  Interventions: Drug: placebo; Drug: Aspirin; Drug: Clopidogrel

INTERVENTIONS:
Drug: tirofiban in PV — a loading dose of 10ug/kg tirofiban is given in 3 min through PV,followed by a maintenance dose of 0.15ug/kg*min for 48h.
  (clopidogrel 600 mg+aspirin( ASA) 300 mg)x1 day.
  Other Names: GPⅡb/Ⅲa receptor antagonist
  Arms: tirofiban in PV
Drug: tirofiban in IC — a loading dose of 10ug/kg tirofiban is given in 3 min through IC,followed by a maintenance dose of 0.15ug/kg*min for 48h.
  (clopidogrel 600 mg+ ASA 300 mg)x1 day.
  Other Names: GP IIb/IIIa receptor antagonist
  Arms: tirofiban in IC
Drug: antiplatelet thrombolysin — a loading dose of 5 IU/60kg in 5 min through PV,followed by a maintenance dose of 0.002 IU/kg/h for 48h.
  (clopidogrel 600 mg+ ASA 300 mg)x1 day.
  Other Names: GP Ib receptor antagonist
  Arms: antiplatelet thrombolysin
Drug: placebo — a loading dose of 5 IU/60kg in 5 min through PV,followed by a maintenance dose of 0.002 IU/kg/h for 48h.
  (clopidogrel 600 mg+ ASA 300 mg)x1 day.
  Arms: placebo
Drug: Clopidogrel — loading dose of 300 mg clopidogrel followed by a maintenance dose of 75 mg/d for at least 5 days
  Arms: dual antiplatelet therapy
Drug: Aspirin — loading dose of 300 mg aspirin followed by a maintenance dose of 100 mg/d for at least 5 days.
Drug: Clopidogrel — loading dose of 600 mg clopidogrel followed by a maintenance dose of 75 mg/d for at least 5 days
  Arms: antiplatelet thrombolysin; placebo; tirofiban in IC; tirofiban in PV

SUMMARY:
Antiplatelet treatment is important for coronary artery disease(CAD) patients .Some patients are resistant to antiplatelet treatment based on platelet function tests(PFT).Currently the results of PFT are mainly based on the analysis of peripheral blood. instead, adverse cardiovascular events in CAD patients may be more directly related to platelet activities in the coronary arteries. There's no evidence of system study to prove the PFT of peripheral blood can represent the platelet functions in coronary arteries.The purpose of this study is to determine the different platelet activities in the blood of peripheral vein (PV), peripheral artery (PA), intracoronary artery (IC) in the CAD patients without or with different interventions.

our study is divided into three parts: Part A: To study the different platelet activities in the blood of PV, PA, IC in the CAD patients with dual antiplatelet therapy.

Part B: To explore the different platelet activities of the above three sites in ST-segment elevation myocardial infarction (STEMI) patients who are administrated platelet membrane glycoprotein Ⅱb/Ⅲa (GPⅡb/Ⅲa) receptor antagonist ( tirofiban ) in PV or IC and dual antiplatelet therapy.

Part C: To explore the different platelet activities of the above three sites in STEMI patients who are administrated antiplatelet thrombolysin or placebo in PV and dual antiplatelet therapy.

DETAILED DESCRIPTION:
Part A:A total of 30 CAD patients are recruited.All patients are on loading dose of 300 mg clopidogrel followed by a maintenance dose of 75 mg/d for at least 5 days and a loading dose of 300 mg aspirin followed by a maintenance dose of 100 mg/d for at least 5 days. All patients plan to receive coronary arteriography (CAG) or percutaneous coronary intervention (PCI).The investigators sample blood from PV,PA and IC before PCI.Regional differences will be compared between blood samples from PV,PA and IC by light aggregometry (agonists: arachidonic acid, LTA-AA; adenosine diphosphat, LTA-ADP), VerifyNow P2Y12 assays. Differences between LTA and VerifyNow P2Y12-assay will also be compared.

Part B:A total of 30 STEMI patients are recruited.Patients are randomly assigned to 2 groups.A group(n=15) is given tirofiban through PV, the other group(n=15) is given through IC.All patients are on loading dose of 600 mg clopidogrel and 300 mg aspirin.All patients plan to receive emergency PCI. Group PV: a loading dose of 10ug/kg tirofiban is given in 3 min through PV,followed by a maintenance dose of 0.15ug/kg*min for 48h.Group IC: a loading dose of 10ug/kg tirofiban is given through IC,followed by a maintenance dose of 0.15ug/kg*min for 48h. Blood samples are collceted from PV, PA and IC before the injection of loading dose tirofiban , and 15min after the injection.Regional differences will be compared between blood samples from PV,PA and IC by LTA-AA; LTA-ADP, LTA-RIS(agonists:ristocetin),VerifyNow P2Y12 assays.

Part C:A total of 30 STEMI patients are recruited.Patients are randomly assigned to 2 groups.A group(n=15) is given antiplatelet thrombolysin(the frist antiplatelet drugs based on GP Ib receptor which completed the preclinical and phase I clinical studies,and already has entered phase II clinical studies) through PV, the other group(n=15) is given placebo through PV.All patients are on loading dose of 600 mg clopidogrel and 300 mg aspirin.All patients plan to receive emergency PCI.Both Groups are given in the same way , a loading dose of 5 IU/60kg in 5 min through PV,followed by a maintenance dose of 0.002 IU/kg/h for 48h. Blood samples are collceted from PV, PA and IC before the injection of loading dose of antiplatelet thrombolysin or placebo, and 15 min after the injection.Regional differences will be compared between blood samples from PV,PA and IC by LTA-AA; LTA-ADP, LTA-RIS and VerifyNow P2Y12 assays.

ELIGIBILITY:
Inclusion Criteria:

1. CAD patients plan to receive coronary arteriography (CAG) or percutaneous coronary intervention (PCI).
2. Patient aged >18 years and ≦75 years old;
3. Signed inform consent

Exclusion Criteria:

1. Allergy or intolerance to ASA, clopidogrel , tirofiban ,antiplatelet thrombolysin;
2. Subjects at a high risk of bleeding (e.g. platelet count< 100*109/L, known bleeding diathesis , active peptic ulcer );
3. Patients who are planning to take warfarin or drugs that potentially could interfere with the anti-platelet effects .
4. severe hemodynamic instability
5. severe liver and renal dysfunction

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
platelet aggregation | 2 hours
  Regional differences between blood samples from PV,PA and IC by LTA and VerifyNow P2Y12 assays.The results of LTA are reported in platelet aggregation rate（%）.Platelet aggregation was induced using 0.5 mg/ml arachidonic acid (AA) and 5 μmol/l ADP.The maximum aggregation achieved during an 8-minute period was used for analysis.The results of the VerifyNow P2Y12-assay are reported in P2Y12 reaction units (PRU).(using 20 μmol/l ADP as the agonist and 22 nmol/l prostag- landin E1 (PGE1). a value that uses iso- thrombin receptor-activating peptide to approximate a baseline off-drug platelet reactivity value, and percentage inhibition.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China